CLINICAL TRIAL: NCT01930305
Title: Effects of Heating Transfusion on Brain Function of Surgical Patients
Brief Title: Effects of Heating Transfusion on Brain Function
Status: Completed | Type: Observational
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NXKJGG2012
Record Dates: First submitted 2013-07-17; First posted 2013-08-28 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Blood Transfusion
Keywords: Heating transfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To inversitage whether routine warming of blood is harmful to brain fuction of sugical patients receiving massive transfusion.

DETAILED DESCRIPTION:
Hypothermia is an effective therapeutic intervention to reduce hypoxic ischemia brain injury in animal experiments and in clinics.In a recent study, it has been shown that perioperative warming was associated with a higher incidence of cognitive dysfunction in elderly patients.Therefore, we hypothesised that perioperative heating transfusion have a side effect on brain function of surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for major surgery under general anesthesia and they probably need a blood transfusion during the procedure.

Exclusion Criteria:•Patients with a history of stroke, central nervous system disease , metabolic disturbance, psychiatric illness, hearing impairment, drug abuse or unwilling to participate in assessment

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult paitents scheduled for major surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Brain fuction during perioperative period | Change from baseline at post-transfusion 15min, 30min, 1hour, 2hour, 3 hour, 6hour, 12hour, 24hour
  Brain function includes cerebral blood flow and cerebral oxygen saturation

SECONDARY OUTCOMES:
the cognitive performance and the score of postoperative quality recovery scales ( PQRS) | Chang from baseline at 15min,40min,1day,3day and 7day postoperative lay

OTHER OUTCOMES:
serum concentration of inflammatory cytokine | change from baseline at 3hour, 6hour, 12hour, 24hour after transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Xinli Ni, Study Director — Ningxia Medical University
Locations (2):
- China (2):
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Ningxia Medical University, Yinchuan, Ningxia